CLINICAL TRIAL: NCT06218095
Title: Investigation of Simulation Teaching Efficiency in Evaluation of Thromboembolism Risk in Pregnancy and Postpartum Period
Brief Title: Pregnancy and Postpartum Period Venous Thromboembolism and Simulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, NURCAN ÇAĞLAYAN, Phd Midwifery, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: PhD Midwifery
Record Dates: First submitted 2023-12-28; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Simulation; Venous Thromboembolism
Keywords: teaching with simulation; venous thromboembolism during pregnancy; postpartum embolism; midwifery student training
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): 3rd grade midwifery students experimental group Diagnostic Information Form and Thromboembolism Information Form were applied before the theory training.
  Pregnancy and postpartum thromboembolism theory training was given,
  1. st application: Deep vein thrombosis management scenario during pregnancy A high-validity simulation scenario was implemented. Student Satisfaction and Self-Confidence Scale in Learning after the application, Simulation Design Scale implemented
  2. nd application: It will be done after 2 weeks. Postpartum Embolism Management Scenario was implemented Student Satisfaction and Self-Confidence Scale in Learning after the application, Simulation Design Scale will be applied. Thromboembolism Information Form - Posttest Done After 2 Weeks After 2 months, Thromboembolism Information Form - Persistence Test was performed.
  Interventions: Other: Simulation application
- control group (No Intervention): 3rd grade midwifery students Control group Diagnostic Information Form and Thromboembolism Information Form were applied before the theory training.
  Thromboembolism Information Form-Posttest was applied 1 month later. After the Last Test, Thromboembolism Information Form - Persistence Test was applied 2 months later.

INTERVENTIONS:
Other: Simulation application — Teaching the risk of thromboembolism during pregnancy and postpartum through simulation
  Arms: Experimental

SUMMARY:
This research will be carried out to determine the effectiveness of teaching thromboembolism risk assessment during pregnancy and postpartum period to midwifery students using a high-tech simulation method.

Thromboembolism during pregnancy and postpartum period is one of the preventable causes of maternal deaths. For this reason, it is important to determine the thromboembolism risk of pregnant women and postpartum women by midwives before complications develop and to plan preventive interventions. The aim of the research is to provide midwifery students with the ability to evaluate the risk of thromboembolism before clinical experience through high-tech simulation application.

Goals;

* To increase midwifery students' skills in assessing thromboembolism risk during pregnancy and postpartum period before clinical practice.
* To increase the self-confidence and satisfaction of midwifery students with simulation application in pregnancy and postpartum thromboembolism risk assessment skills.
* To develop midwifery students' quick, critical thinking and decision-making skills in assessing the risk of thromboembolism before clinical practice.
* To help midwifery students visualize the risk of pregnancy and postpartum thromboembolism, which has an important place in terms of maternal deaths, by creating a clinical environment with a case scenario.
* To determine the effectiveness of midwifery teaching through case scenario simulation application with the risk of pregnancy and postpartum thromboembolism, and to increase students' learning and clinical practice skills.

DETAILED DESCRIPTION:
Design of the Research: Researchers will receive scenario creation and simulation design training for the advanced technology simulation method. After the simulation training, pregnancy and postpartum thromboembolism scenarios will be prepared for the intervention group. A thromboembolism information form will be prepared for the intervention and control groups. Expert opinions will be obtained from at least 6 people who are experts in the field of risky pregnancy and postpartum on the forms and scenarios prepared by the researcher. In line with expert opinions, the scenarios and thromboembolism information form will be finalized. The scenarios and forms prepared for the intervention group will be piloted with 6 3rd year midwifery students and volunteers, and final corrections will be made.

Two groups, the intervention and control groups, will be given a 2-hour theoretical training on the risks of pregnancy and postpartum thromboembolism prepared by the researchers. Then, the "Thromboembolism information evaluation form" will be applied to the intervention and control groups. The control group will not be taught with the simulation method.

After the pilot application, the intervention group will be given a laboratory environment close to the clinical environment and will be given scenarios prepared with simulation method teaching and thromboembolism risk assessment training. The simulation application teaching period is planned to be 45 minutes in total, with the first 10 minutes of preliminary information, 15 minutes of teaching with the simulation method, and the last 20 analysis sessions. Afterwards, the thoughts of each 6 students regarding simulation training and teaching will be evaluated in the analysis sessions. Then, the thromboembolism information form and the two scales to be used will be applied to the Intervention group. It is planned to apply the same application to the intervention group twice in total, with an interval of 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Having a statement of consent
* Being a third year midwifery student
* Having taken the risky pregnancy and birth course

Exclusion Criteria:

* Wishing to withdraw from the research at any time.
* Not participating in all simulation applications
* Incompletely filling out data collection forms

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-08-10 (Estimated)

PRIMARY OUTCOMES:
Thromboembolism Information Sheet | Thromboembolism Information Form - is applied 3 times within 3 months as pre-test, post-test and permanence.
  Thromboembolism Information Sheet,Thromboembolism Information Form is a three-part form consisting of 20 questions. Each question is worth 5 points. (Max:100, Min:0)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Midwifery Simulation Laboratory, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data will be shared 6 months after publication.